CLINICAL TRIAL: NCT00259233
Title: The Effects of Peripheral Administration of Saline, PYY1-36 and PYY3-36 on ad Libitum Energy Intake and Appetite.
Brief Title: The Role of Peptide YY (PYY)in Inhibiting Food Intake.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Aditech Pharma AB (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: B208, 2
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2007-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Drug: peripheral Peptide YY administration

SUMMARY:
12 obese subjects will receive peripheral administration of placebo and 4 escalating doses of PYY1-36 and another 12 obese subjects will receive peripheral administration of placebo and 4 escalating doses PYY3-36 on 5 different test days within one week. The patients will be tested in a single blinded dose escalating protocol. Measurements of appetite, ad libitum energy intake, blood pressure and blood sampling will be performed during the test day.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (BMI: 18-23 kg/m2) or 12 overweight/obese (BMI: 27-40 kg/m2)
* Body weight fluctuations < 5 kg over the past 2 months.
* Blood pressure normal to mildly hypertensive(<159/99 mm Hg)
* Non-elite athletes and not planning to change physical activity during the study.

Exclusion Criteria:

* Any physiological or psychological illnesses that could influence the study results.
* Regular use of medicine.
* Smoking defined as <1 cigarette per day.
* Substance abuse or dependence.
* Blood donation within the past 3 months before entering the study.
* Drinking >21 alcoholic units/week.
* Food allergies.
* Special diets (e.g. vegetarian) or dislikes to any of the foods served during the study.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2005-03; Study Completion 2005-05

PRIMARY OUTCOMES:
appetite
energy intake

SECONDARY OUTCOMES:
Plasma PYY profile
Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor, Principal Investigator — Department of Human Nutrition, RVAU